CLINICAL TRIAL: NCT06728371
Title: Intravenous Methadone for Sternotomy Pain Control in Cardiac Surgery: Double-blinded, Randomized Controlled Trial
Brief Title: Intravenous Methadone for Sternotomy Pain Control in Cardiac Surgery
Acronym: MethadoneRCT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, WONG MAN KIN, Principal Investigator, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CUHK_PWH
Record Dates: First submitted 2024-11-28; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Methadone; Morphine

STUDY DESIGN:
Intervention Model Description: Single centred, parallel, double blinded, randomized controlled trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: By drawing sequentially numbered, coded sealed, opaque envelops each containing the group assignment of either methadone or morphine group. The sealed envelopes for randomization will be prepared by a third party who takes no further part in the study. The study syringes containing the drug solution will be prepared by a nurse not involved in the study with blind labelling. The primary care team, blinded to the group allocation, will perform all surgical procedures using standardized techniques. Anaesthetists and nurses blinded to group allocation will record data intraoperatively, in ICU, and at regular intervals in the cardiac wards.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Methadone group: Intervention (Experimental): 0.2mg/kg methadone
  Interventions: Drug: Methadone
- Morphine group: control (Active Comparator): Equipotent dose of morphine (0.2mg/kg)
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Methadone — 0.2mg/kg intravenous methadone given at induction
  Other Names: Methadone: Intervention
  Arms: Methadone group: Intervention
Drug: Morphine — 0.2mg/kg intravenous morphine given at induction
  Other Names: Morphine: control
  Arms: Morphine group: control

SUMMARY:
Background Postoperative pain is significant in cardiac surgical patients. Perioperative analgesia with intermittent administration of opioids can result in significant fluctuations in serum opioid concentrations. Methadone should provide a rapid onset and long-term pain relief upon a single intravenous dose at induction of anaesthesia, and may reduce chronic postsurgical pain (CPSP) in cardiac surgical patients. The feasibility of using intravenous methadone in Chinese cardiac surgical patients, and its effect on acute and chronic pain management after cardiac surgery will be evaluated.

Methods A single-centre, prospective, randomized-controlled study. Adult cardiac surgical patients will be randomized to receive either methadone 0.2mg/kg (maximum dose 20mg) or equipotent dose of morphine at induction of anaesthesia. Patient-controlled analgesia morphine protocol, oral paracetamol and dihydrocodeine will be given for postoperative analgesia. Venous blood sampling for plasma methadone concentration will be obtained at regular intervals from study drug infusion to 96 hours after administration. The primary outcomes will be the recruitment and attrition rate, complications from methadone, and the perceived trial feasibility. Secondary outcomes include time weaned to spontaneous breathing trial, morphine consumption within 24 hours and 72 hours after surgery, time to first morphine rescue, postoperative pain score, patient satisfaction, length of stay in ICU and hospital. Side effects of opioids including sedation, nausea and vomiting, and time to first bowel opening will be recorded. CPSP will be assessed with DN4 questionnaire at 3 and 6 months after surgery.

DETAILED DESCRIPTION:
PAIN IN CARDIAC SURGERY Despite modern day improvements in pain treatment and availability of different analgesic modalities, suboptimal postoperative pain control remains an issue in cardiac surgical patients. Acute postoperative pain is common among cardiac surgical patients, particularly within the first 2 days after surgery, with reported at least moderate intensity. There could be many facets for postoperative pain after adult cardiac surgery. Pain can be caused by surgical incisions and dissections, sternal fracture or incomplete bone healing, multiple drainage cannulas and chest tubes and sternal wound infections. Poorly controlled acute postoperative pain is associated with adverse physiological outcomes that impair the recovery of cardiac surgical patients. It is associated with decreased patient satisfaction, delayed postoperative ambulation, and the development of chronic postsurgical pain (CPSP). The association between sternotomy pain and pulmonary complications has been observed, and the sympathetic activation secondary to pain can induce myocardial ischemia and arrhythmias. Pain control has also been pointed out as one of the major concerns to cardiac surgical patients in intensive care unit. Therefore, optimal acute pain control not only can improve clinical outcomes, but also improves patient satisfaction after cardiac surgery.

Postoperative pain that persists beyond the normal time for tissue healing is increasingly recognized as an important complication after various types of surgery. According to the International Association for Study of Pain, CPSP is defined as the persistence of pain at surgical site or referred area, at least 3 months following the surgical procedure. CPSP is common after cardiac surgery. The reported incidence was 28% to 56% up to 2 years postoperatively. Several mechanisms have been involved in the development of chronic pain after sternotomy. These include dissection, nerve entrapment by sternal wires, sternal retraction, ribs fractures, and intercostal neuralgia as a consequence of nerve damage during dissection of the internal mammary artery during coronary artery bypass graft (CABG). In addition, poorly controlled pain has been a general risk factor for the development of CPSP. All can stimulate the release of pro-inflammatory cytokines which sensitize the afferent nociceptive fibres to cause chronic pain. CPSP has the potential to impact daily functioning and quality of life of patients, as well as increasing the healthcare costs. CARDpain study reported that among those with CPSP, over 50% had significant pain-related interferences with activities of daily living (family and home responsibilities, recreation and employment) at 3, 6 and 12 months following cardiac surgery. Therefore, apart from optimal acute pain control, it is equally important to prevent and manage CPSP, to ensure better satisfaction and quality of lives for our patients.

CHALLENGES IN PAIN MANAGEMENT Intravenous opioids such as fentanyl and morphine have been the mainstay of perioperative analgesia for cardiac surgery, either by intermittent boluses or through a patient-controlled device. The primary problem with this mechanism of delivery is that significant fluctuations in serum opioid concentrations can occur, resulting in effects which range from inadequate analgesia to overdose and respiratory depression. These peaks and troughs of analgesia that occur with intermittent opioids administration may explain the suboptimal pain control during the initial postoperative period. In contrast to intermittent administration of short-acting opioids such as morphine and fentanyl, a single dose administration of methadone can be considered. Methadone was conventionally used in cancer and chronic pain management. It can be administered via oral, intravenous, and other parenteral routes. Despite being an often-used alternative to morphine, it remains relatively invisible in perioperative settings. Methadone is a unique opioid that may provide several important potential benefits for surgical patients in the perioperative period. It is a potent mu receptor agonist with a rapid onset and longest half-life (24-36 hours) of the clinically used opioids. According to a pharmacokinetic study, central nervous system effect site methadone concentration rapidly equilibrates with plasma concentrations, evidenced by a short lag time between plasma concentrations and effects (t1/2ke0 4min). This is comparable to the rapid onset and effect compartment equilibration of fentanyl and sulfentanil (5-6min), and in contrast the slow onset time of morphine, where t1/2ke0 has been reported to exceed 4 hours. In addition, as reviewed in an editorial, when methadone is administered at a dose of 20mg or higher, the duration of analgesia approximates the half-life of 24-36 hours. Therefore, a single intravenous dose 20mg administered to an adult at induction of anaesthesia should provide a rapid onset and significant pain relief up to 1-2 days postoperatively, which is the period reported to have the highest pain score after cardiac surgery. Methadone is also a N-methyl-D-aspartate (NMDA) receptor antagonist. It has been reported to possess anti-hyperanalgesic and anti-allodynic properties, that is important in preventing pain sensitization and the development of CPSP, which is of high risk in cardiac surgical patients.

SIDE EFFECTS OF METHADONE Methadone shares the same opioid-related side effects as with many other opioids such as nausea and vomiting, drowsiness and respiratory depression. According to a meta-analysis in 2020 which included seven randomized controlled trials on intraoperative use of intravenous methadone, four studies reported no adverse events. One study reported that the patients who received intraoperative methadone experienced more sedation compared to control group at 24 hours after surgery. One study reported that the intraoperative morphine group had more sedation compared to methadone group during the postoperative period. Methadone was not shown to have a higher incidence of postoperative nausea and vomiting compared to the morphine group. Methadone has been reported to be associated with cardiac conduction abnormalities such as QT prolongation, QT interval dispersion and cardiotoxicity (Torsade de pointes). However, most of the cardiac-related side effects were seen in patients on prolonged or maintenance treatment with methadone. Significant dose-dependent QTc prolongation usually occurs at a high dose of methadone. A single injection of intravenous methadone at low dose is unlikely to result in significant cardiotoxicity. No cardiac disturbances were reported from the meta-analysis.

GAPS IN THE LITERATURES Only a few trials have studied intravenous methadone as an analgesic in surgical patients, in particular, there have not been many studies in the field of cardiac anaesthesia. A randomized controlled trial done by Murphy et al showed intraoperative methadone to be superior to fentanyl for patients undergoing cardiac surgery. Methadone was demonstrated to reduce morphine consumption in the first 24 postoperative hours and improved pain scores at 12h after extubation compared to patients receiving fentanyl. There was 40% reduction in morphine requirement during the first 24h after extubation, and the severity of postoperative pain was decreased by 30-40% during the first three days after cardiac surgery. There was only one study comparing the analgesic efficacy between methadone and morphine give at the time of induction in cardiac surgical patients. Methadone was shown to reduce opioid requirement at 24h postoperatively and significantly reduce the incidence of postoperative nausea and vomiting. So far there has not been any studies on using methadone for cardiac surgery in Chinese populations, and none on the role of methadone for prevention of chronic post-surgical pain in cardiac surgical patients. Substantial literatures have demonstrated the ethnic differences in pain perception and endogenous pain modulation is postulated to be a mechanism for ethnic differences. Studies comparing Caucasians and Asians, such as Chinese and Indians, generally demonstrated lower pain tolerance in Asian populations. The primary aim of this pilot trial is a feasibility study to evaluate the protocol and the effect of methadone on acute and chronic pain control after open cardiac surgery, compared with conventional opioid-based approach using morphine and fentanyl. In addition, the effects of methadone on opioids consumption, opioid-related side effects, patient satisfaction, postoperative extubation times, and length of stay in hospital and ICU will be determined.

Randomization and concealment Patients will be randomized to receive either methadone 0.2mg/kg (maximum dose 20mg) or equipotent dose of morphine, adding to a syringe containing saline made up to 50ml in total, by drawing sequentially numbered, coded sealed, opaque envelops each containing the group assignment of either methadone or morphine group. The sealed envelopes for randomization will be prepared by a third party who takes no further part in the study. The study syringes containing the drug solution will be prepared by a nurse not involved in the study with blind labelling. The primary care team, blinded to the group allocation, will perform all surgical procedures using standardized techniques. Anaesthetists and nurses blinded to group allocation will record data intraoperatively, in ICU, and at regular intervals in the cardiac wards.

Eligibility criteria We will include adult patients age 18 or older, undergoing elective coronary artery bypass graft (CABG), valve repair/replacement, or combined CABG/valve procedure via sternotomy, with an expected extubation within 12 hours of surgery. The exclusion criteria include emergency surgery, aortic surgery, redo surgery, preoperative renal failure requiring renal replacement therapy or creatinine clearance <30ml/min (calculated by Cockcroft-Gault formula), liver dysfunction (liver enzymes twice upper limit normal), LVEF <40%, requirement of mechanical hemodynamic support in perioperative period, history of chronic pain or who regularly used pain medications (except paracetamol and non-steroidal anti-inflammatory drugs), history of psychiatric illnesses or illicit drug use, intraoperative use of remifentanil and unable to provide informed consent.

Anaesthesia and interventions All patients will receive standard monitoring for cardiac surgery. General anaesthesia will be induced with midazolam 0.01-0.05mg/kg, fentanyl 2-5mcg/kg and rocuronium 0.5-1mg/kg to facilitate intubation with single-lumen cuffed endotracheal tube. Anaesthesia will be maintained with sevoflurane and propofol infusion that target Bispectral Index 40-60. The study drug (either methadone 0.2mg/kg or morphine at equipotent dose) in blind labelling will be administered at time of induction by intravenous infusion over 30 minutes. No further morphine will be given throughout the operation. No other analgesics (paracetamol, non-steroidal anti-inflammatory agents, dexmedetomidine, ketamine), steroids or antiemetics will be given intraoperatively. Patient-controlled analgesia (PCA) morphine protocol will be prescribed to patients for 72 hours after operation for postoperative analgesia. Oral analgesics including paracetamol 1g every 6 hours and dihydrocodeine 30mg three times a day will be prescribed by parent surgical team. At the end of the operation, the patients will be kept sedated with propofol infusion to ICU. Propofol infusion will be stopped upon admission to ICU to facilitate weaning from ventilator. Adaptive Support Ventilation (ASV) is used in ICU for weaning which adjusts the ventilation parameters depending on the patient's lung mechanics and effort. Pain will be assessed by nurses in ICU at 4h after stopping sedation, then once every 2h. Upon extubation, patient will be assessed the pain score and the level of sedation at 15min, 8h, 12h, 24h, 48h and 72h. 1mg morphine will be administered via PCA to patients if pain of more than mild severity was noted. Any nausea or vomiting, and use of rescue antiemetics will be documented.

ELIGIBILITY:
Inclusion Criteria:

* adult patients age 18 or older
* elective coronary artery bypass graft (CABG), valve repair/replacement, or combined CABG/valve procedure via sternotomy
* Expected extubation within 12 hours of surgery.

Exclusion Criteria:

* emergency surgery
* aortic surgery
* redo surgery
* preoperative renal failure requiring renal replacement therapy or creatinine clearance <30ml/min (calculated by Cockcroft-Gault formula)
* liver dysfunction (liver enzymes twice upper limit normal)
* LVEF <40%
* mechanical hemodynamic support in perioperative period
* history of chronic pain or who regularly used pain medications (except paracetamol and non-steroidal anti-inflammatory drugs)
* history of psychiatric illnesses or illicit drug use
* intraoperative use of remifentanil
* unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative morphine consumption | Postoperative within 72 hours
  Morphine consumption within 72h postoperative time frame

SECONDARY OUTCOMES:
Pain score | Within 72 hours postop
  Measured using Numerical Rating Scale. It ranges from 0-10. The higher the score, the worse the pain
Time to first morphine rescue | from immediately after the operation till Day 1
  time the patient feels the need to use morphine from patient-controlled analgesia machine
ventilator time | from immediately after the operation till Day 1
  The time at which the patient successfully weaned to spontaneous breathing according to ICU ASV protocol
Nausea and vomiting | postoperatively within 72 hours
  Number of episodes of postoperative nausea and vomiting
Length of hospital stay | up to 1 month after surgery
  Number of hours the patient spent in hospital
Length of ICU stay | up to 1 week after surgery
  Number of hours the patient spent in ICU
Chronic postsurgical pain at 3 months | Measured at 3 months after surgery
  Measured using Douleur Neuropathique en 4 questionnaire. It ranges from 0 to 10. A score greater than or equal to 4 indicates the diagnosis of chronic pain
Chronic postsurgical pain at 6 months | Measured at 6 months after surgery
  Measured using Douleur Neuropathique en 4 questionnaire. It ranges from 0 to 10. A score greater than or equal to 4 indicates the diagnosis of chronic pain

CONTACTS AND LOCATIONS:
Overall Officials: Man Kin Wong, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

DOCUMENTS (2):
  • Study Protocol: Study protocol (2024-11-28): https://cdn.clinicaltrials.gov/large-docs/71/NCT06728371/Prot_000.pdf
  • Informed Consent Form (2024-11-28): https://cdn.clinicaltrials.gov/large-docs/71/NCT06728371/ICF_001.pdf